CLINICAL TRIAL: NCT04340895
Title: Pragmatic Randomized Controlled Study to Assess the Effectiveness of Two Patient Management Strategies in Mild to Moderate Ulcerative Colitis
Brief Title: Study to Assess Effectiveness of Therapy Timely Adjustment Based on Self-monitoring in Patients Suffering From Mild-to-moderate Ulcerative Colitis (OPTIMISE Study)
Acronym: OPTIMISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 7002661
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Mild-to-moderate Ulcerative Colitis
Keywords: Ulcerative Colitis; Management strategies; Pragmatic trial
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Treatment optimization (escalation/de-escalation) performed by the investigator based on participant self-monitoring of FC values and/or clinical symptoms (patient-reported outcome-2 [PRO-2] scoring).
  The FC Test and/or PRO-2 scoring will be done by the participant at home every month during active disease, every 3 months in remission, or when a participant feels the need/presents clinical symptoms.
  Interventions: Other: Faecal Calprotectin Home Test; Other: PRO-2 Scoring
- Reference arm (Active Comparator): Treatment optimization (escalation/de-escalation) performed by the investigator based on clinical symptoms (PRO-2 scoring) only.
  The PRO-2 scoring will be assessed during clinic visits every 3-months during active disease, every 6 months during remission, or when a participant feels the need; as per recommended standard practice.
  Interventions: Other: PRO-2 Scoring

INTERVENTIONS:
Other: Faecal Calprotectin Home Test — A non-invasive, in vitro diagnostic test for the determination of FC levels in human stool samples in combination with the dedicated 'CalproSmart' smartphone application.
  This test helps participants to self-monitor their FC levels at their own homes, ensuring an adequate and effective medical treatment regimen performed by the investigator.
  Arms: Intervention arm
Other: PRO-2 Scoring — Monitoring of clinical symptoms will be performed by PRO-2 scoring, which includes rectal bleeding (RB) and stool frequency (SF) assessment obtained within the last 3-days.

SUMMARY:
The purpose of this study is to provide evidence that a therapy of Ulcerative Colitis (UC) disease adjusted on tight monitoring of non-invasive parameters, such as clinical symptoms and faecal calprotectin (FC) (substance that is released when intestines are inflamed and that can be measured in faeces), can provide significantly higher benefit for the participants in terms of disease control and quality of life (QoL) improvement, compared to a symptom-based approach only.

ELIGIBILITY:
Inclusion Criteria:

* Adult Participants (≥ 18 years old)
* Participants with active mild-to-moderate UC (with RB and bowel inflammation confirmed by endoscopy)
* Participants with treatment with 5-aminosalicylic acid (5-ASA) ≤ 2.4 g/day or with no treatment regimen at Baseline
* Participants who agree to use FC home test (to dose FC in faeces as a marker of inflammation)
* Participants with internet access and smartphone with camera

Exclusion Criteria:

* Participants currently enrolled in another interventional study
* Participants not willing to undergo an endoscopy at the end of study
* Participants with contraindications to treatment with 5-ASA and/or 2nd generation corticosteroids
* Participants not willing to perform FC self-testing in faeces at home

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Mayo Endoscopic Sub-score = 0 | At 12 months
  Defined as the percentage of participants achieved mucosal healing (Mayo endoscopic sub-score of 0 [normal friability]). The Mayo endoscopic scoring ranges from 0-3 with higher scores indicating greater disease severity. The score is defined as 0-3: 0= Normal; 1=Mild friability; 2 = Moderate friability; 3 = Exudation, spontaneous hemorrhage.

SECONDARY OUTCOMES:
Percentage of Participants with Rectal Bleeding = 0 | At 12 months
  Defined as the percentage of participants with no RB (RB=0). The RB score ranges from 0-3 with higher scores indicating greater disease severity. The score was defined as 0-3: 0 = None; 1 = Streak of blood; 2 = Obvious blood; 3 = Mostly blood
Percentage of Participants with Stool Frequency <=1 | At 12 months
  Defined as the percentage of participants with SF<=1. The SF score ranges from 0-3 with higher scores indicating greater disease severity. The score was defined as 0-3: 0 = None; 1 = 1-2 stools/day > normal; 2 = 3-4 stools/day > normal; 3 = >4 stools/day > normal
Percentage of Participants with Mayo Endoscopic Sub-score <=1 | At 12 months
  Defined as the percentage of participants achieved endoscopic remission (Mayo endoscopic sub-score <=1 [normal or mild friability]). The Mayo endoscopic scoring ranges from 0-3 with higher scores indicating greater disease severity. The sub-score was defined as 0-3: 0 = Normal friability; 1 = Mild friability; 2 = Moderate friability; 3 = Exudation, spontaneous hemorrhage
Change in Short Inflammatory Bowel Disease Questionnaire (SIBDQ) | From Baseline over 12 Months
  Defined as a change in the QoL using SIBDQ over 12 months. The SIBDQ consists of 10 questions, measuring systemic, social, Bowel, and emotional status; each question is scored on a scale from 1 (poor QoL) to 7 (optimum QoL). A higher score indicates a better QoL. Total scores range from 10 (poor QoL) to 70 (good QoL).
Change in Short Form Questionnaire-36 (SF-36) | From Baseline over 12 Months
  The SF-36 is a health-related survey that assesses participant's QoL and consists of 36 questions covering 8 health domains: physical functioning, bodily pain, role limitations due to physical problems and emotional problems, general health, mental health, social functioning, vitality, and 2 component scores (mental component score and physical component score). Each domain is scored by summing the individual items and transforming the scores into a 0 (poorest health) to 100 (best health) scale with higher scores indicating better health status or functioning.
Percentage of Participants Escalated to Rescue Therapy | Over 12 months
  Rescue therapy included systemic corticosteroids/ immunosuppressants /biologics.
Change in Work Productivity and Activity Impairment: Ulcerative Colitis (WPAI: UC) Questionnaire | From Baseline over 12 Months
  The WPAI-UC is a questionnaire with 6 questions used to evaluate lost productivity (work time missed and work and activity impairment) during the past 7 days due to UC. The scores are presented as percentages.
Number of Hospitalization Days | Over 12 months
  Number of hospitalization days will be determined by UC related medical resources.
Number of Outpatients Visits and Calls (Outside of Study Schedule) | Over 12 months
  Number of outpatients visits and calls (outside of study schedule) will be determined by UC related medical resources.
Number of Ulcerative Colitis Related Procedures and/or Surgeries | Over 12 months
  Number of UC related procedures and/or surgeries will be determined by UC related medical resources.
Faecal Calprotectin Value Changes at the Defined Study Time Points (Interventional Arm Only) | Over 12 months
  The FC Test will be done by the participant at home every month during active disease, every 3 months in remission, or when participant feels the need/presents clinical symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (42):
- Czechia (6):
  - Vojenska nemocnice Brno p.o., Brno
  - Hepato-Gastroenterologie HK, s.r.o., Hradec Králové
  - EGK s.r.o. - Sanatorium sv. Anny, Prague
  - ISCARE IVF a.s., Prague
  - Mediendo s.r.o., Prague
  - KZ a.s. - Masaryk Hospital, Ústí nad Labem
- Hungary (7):
  - Semmelweis Egyetem, Isz. Sebeszeti es Intervencios Gasztroenterologiai Klinika, Budapest
  - Pannonia Mgánorvosi Centrum Kft, Budapest
  - Bugat Pal Hospital, Gyöngyös
  - Bacs-Kiskun Megyei Oktatokorhaz, Kecskemét
  - University of Pecs, Pécs
  - Szegedi Tudomnyegyetem, Szeged
  - Javorszky Odon Hospital, Vác
- Italy (6):
  - AOU Ospedali Riuniti di Ancona, Ancona
  - ASST-FBF Luigi Sacco Hospital, Milan
  - Ospedale San Raffaele S.R.L, Milan
  - Ospedali Riuniti Villa Sofia-Cervello, Palermo
  - Azienda Ospedaliero - Universitaria Pisana, Pisa
  - A.O.Città della salute e della scienza diTorino, Torino
- Netherlands (3):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Catharina Ziekenhuis, Eindhoven
  - Franciscus Gasthuis & Vlietland, Rotterdam
- Poland (16):
  - NZOZ Vitamed, Bydgoszcz
  - Szpital Uniwersytecki, Bydgoszcz
  - Osrodek Sadan Klinicznych CLINSANTE, Bydgoszcz
  - Centrum Medyczne LukaMed, Chojnice
  - Karkonoskie Centrum Bada Klinicznych - Lexmedica SP Z O O, Jelenia Góra
  - Centrum Medyczne Promed, Krakow
  - SANTA FAMILIA Centrum Badan Profilaktyki i Leczenia, Lodz
  - Orodek Bada Klinicznych Allmedica, Nowy Targ
  - Centrum Medyczne Medyk, Rzeszów
  - Korczowski Bartosz, Gabinet Lekarski, Rzeszów
  - H-T. Centrum Medyczne sp. z o.o., Tychy
  - Centralny Szpital Kliniczny Ministerstwa Spraw, Warsaw
  - NZOZ Centrum Gastroenterologii w Wodzislawiu Slaskim, Wodzisław Śląski
  - Melita Medical, Wroclaw
  - Centrum Diagnostyczno Lecznicze Barska, Włocławek
  - Clinhouse Centrum Medyczne, Zabrze
- Slovakia (4):
  - ENDOMED s.r.o., Košice
  - Pigeas s.r.o., Martin
  - Fakuktna Nemocnica Nitra, Nitra
  - Gastro LM s.r.o., Prešov

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Danese S, Fiorino G, Vicaut E, Paridaens K, Ugur A, Clark B, Vanasek T, Stepek D, D'Amico F, West R, Gilissen LPL, Wisniewska Jarosinka M, Drobinski P, Fronik G, Fic M, Walczak M, Kowalski M, Korczowski B, Wiatr M, Peyrin-Biroulet L. Clinical Trial: A Pragmatic Randomised Controlled Study to Assess the Effectiveness of Two Patient Management Strategies in Mild to Moderate Ulcerative Colitis-The OPTIMISE Study. J Clin Med. 2024 Aug 30;13(17):5147. doi: 10.3390/jcm13175147. PMID 39274360
- [Derived] Dal Buono A, Roda G, Argollo M, Paridaens K, Peyrin-Biroulet L, Danese S. 'Treat to Target' in Mild to Moderate Ulcerative Colitis: Evidence to Support this Strategy. Curr Drug Targets. 2021;22(1):117-125. doi: 10.2174/1389450121666200727120305. PMID 32718289